CLINICAL TRIAL: NCT07214857
Title: Potential Eligibility and Estimated Preventable Cardiovascular Disease Events From Inclisiran Treatment in the United States
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839D1US03
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Disease
Keywords: Prevention; Inclisiran; Statins; Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Secondary Prevention Population: Patients with known ASCVD who met the secondary prevention population eligibility criteria.
- High-risk Primary Prevention Population: Patients without known ASCVD who met the high-risk primary prevention population eligibility criteria.
- Diabetes Population: Patients with diabetes who met the diabetes population eligibility criteria.

SUMMARY:
The aim of this study was to estimate the number of United States (US) adults with and without prior atherosclerotic cardiovascular disease (ASCVD) and diabetes who may be eligible for inclisiran based on US National Health and Nutrition Examination Survey (NHANES) data and inclisiran eligibility criteria from ongoing clinical trials as well as to estimate the number of preventable ASCVD events based on expected risk reductions from the degree of low-density lipoprotein cholesterol (LDL-C) lowering expected from inclisiran.

This study used data from the US NHANES 2011-2020 surveys. NHANES is a national survey which collects medical history, laboratory, and medication information from participants of all ages.

ELIGIBILITY:
Inclusion criteria:

* Aged 18 years of age or older
* Elevated LDL-C despite statin therapy
* Other inclusion criteria per ongoing inclisiran clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a cross-sectional, non-interventional cohort study.
Sampling Method: Probability Sample
Enrollment: 1385 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Estimated Number of US Patients Eligible for Inclisiran Treatment | 10 years
Estimated Number of Preventable Cardiovascular Events Over 10-years of Inclisiran Treatment | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States